CLINICAL TRIAL: NCT05658354
Title: Cognitive Rehabilitation in People With Metabolic Syndrome and Mild Cognitive Deficits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Myrto Koutsonida, PhD candidate, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 27819
Record Dates: First submitted 2022-12-08; First posted 2022-12-20 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Metabolic Syndrome; Cognitive Deficit
Keywords: metabolic syndrome; mild cognitive deficits; computerized cognitive rehabilitation
MeSH Terms: conditions — Metabolic Syndrome; Cognition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computerized cognitive program (Experimental): 25 participants with metabolic syndrome and mild cognitive deficits; receive health advice using the World Health Organization's guidelines for Risk Reduction of Cognitive Decline and Dementia, and perform the computerized cognitive training program (BrainHQ) for 45 minutes per session, twice per week, over the 3-month intervention period.
  Interventions: Other: Computerized cognitive program
- Control group (No Intervention): 25 participants with metabolic syndrome and mild cognitive deficits; receive health advice using the World Health Organization's guidelines for Risk Reduction of Cognitive Decline and Dementia.

INTERVENTIONS:
Other: Computerized cognitive program — BrainHQ was developed by Posit Science and includes computer-based brain-training exercises organized into six categories: Attention, Brain Speed, Memory, People Skills, Intelligence, and Navigation. Participants were instructed to perform a total of 24 sessions of computerized cognitive training at home, consisting of 45 minutes of training, twice per week, over a 3-month period.
  Arms: Computerized cognitive program

SUMMARY:
The goal of this clinical trial is to investigate the possibility of rehabilitation of mild cognitive deficits in people with metabolic syndrome. We aim to implement a cognitive training program on patients with metabolic syndrome and cognitive deficits, and examine its effectiveness both post-intervention (3 months) and after 12 months.

Researchers will compare two groups, the experimental group that will receive the computerized cognitive training and the control group that will receive no training.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Presence of metabolic syndrome according to the criteria of IDF (2005) or revised NCEP-ATP III (2005)
* Presence of mild cognitive deficit (-1.5 SD below age and education-adjusted normative mean) in previously administered neuropsychological tests of Trail Making test (Part A & B), Verbal Fluency test (animals and letter "x"), Logical Memory test (immediate and delayed recall)
* Written informed consent to participate

Exclusion Criteria:

* Presence of any serious neurological or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Change in scores of the Montreal Cognitive Assessment (MoCA) test | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  MoCA is a screening test for mild cognitive dysfunction; range 0-30, higher scores represent better cognitive function
Change in scores of Complex Figure tests | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  Complex Figures assess visuo-constructional ability and visual memory; range 0-36, higher scores represent better cognitive function
Change in scores of Hopkins Verbal Learning Test-Revised (HVLT-R) | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  HVLT-R assesses verbal memory using a list of words; range 0-36 (immediate recall) and range 0-12 (delayed recall), higher scores represent better cognitive function
Change in scores of Digit Span test | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  Digit Span assesses working memory; range 0-14 (performance) and range 2-9 (span) for forward and backward condition, higher scores represent better cognitive function
Change in scores of semantic Verbal Fluency test | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  Verbal Fluency assesses executive function that also relies on language component; higher scores represent better cognitive function
Change in scores of Flanker task | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  Flanker task assesses executive function and inhibition; range 0-48, higher scores represent better cognitive function
Change in scores of Continuous Performance Test (CPT) | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  CPT assesses executive function and inhibition; range 0-100, higher scores represent better cognitive function
Change in scores of Set Shifting | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  Set Shifting assesses executive function and set-shifting; range 0-104, higher scores represent better cognitive function
Change in scores of N-back | baseline, post-intervention (3 months), follow-up (1 year from baseline)
  N-back assesses working memory; range 0-30, higher scores represent better cognitive function

SECONDARY OUTCOMES:
Change in scores of Everyday Cognition-II (Ecog-II) | baseline, follow-up (1 year from baseline)
  Ecog-II is a measure of everyday functioning that includes 41 items to assess memory, language, visual, spatial and perceptual abilities, planning, organization, and divided attention; higher scores represent worse everyday functioning

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hygiene and Epidemiology, School of Medicine, University of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: No